CLINICAL TRIAL: NCT07024368
Title: Reliability of the Sensory Organization Test Over Clinical Administration Time Intervals of Concussion Assessment
Brief Title: Reliability of the SOT Over Clinical Administration Time Intervals of Concussion Assessment
Status: Completed | Type: Observational
Sponsor: Hyung Rock Lee (Other)
Responsible Party: Sponsor-Investigator, Hyung Rock Lee, Associate professor, University of Central Arkansas
Organization: University of Central Arkansas (Other)
Other Study IDs: UGA 2009-10347-5
Record Dates: First submitted 2025-03-18; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-04

CONDITIONS: Healthy; Concussion (Diagnosis); Balance Assessment
MeSH Terms: conditions — Brain Concussion; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Test-retest reliability of the Sensory Organization Test across clinically relevant time intervals: Participants were randomly assigned to one of two groups. Those in the block group completed the SOT following the manufacturer's recommended order, progressing in difficulty from Condition 1 to Condition 6. Those in the random group completed the SOT with conditions presented in a randomized order, generated using MS Excel software.
  These groups will be tested at clinically relevant time intervals: baseline (three tests), Day 45 (follow-up), and Day 50 (additional follow-up).
  Interventions: Device: Reliability of the Sensory Organization Test on the SMART Balance Master across multiple administrations

INTERVENTIONS:
Device: Reliability of the Sensory Organization Test on the SMART Balance Master across multiple administrations — The Sensory Organization Test (SOT) on the SMART Balance Master® will be administered a total of five times. On the first day, participants will complete three SOT sessions, each separated by a 20-minute break. An additional SOT will be conducted on day 45, followed by a final SOT on day 50.
  SOT test scores will be analyzed using Equilibrium Scores (ESs), which provide information on the integration of multiple sensory systems involved in balance through a linear measurement method. Additionally, scores will be evaluated using Multiscale Entropy (MSE), a non-linear model for assessing complexity in postural stability.

SUMMARY:
The goal of this study has two parts. First, it examines whether performing multiple Sensory Organization Tests (SOT) on the SMART Balance Master, using two different testing orders, leads to different levels of practice effects-meaning improvements in balance scores with repeated testing. Second, the study evaluates how reliable the SOT is over time by using two different postural stability measures and two different testing orders. The testing schedule follows the same time intervals commonly used in pre- and post-concussion assessments.

The main hypothesis is that the order of testing-whether done in a blocked or random sequence-affects practice effects on composite and sub-composite balance scores over five repeated SOT sessions.

The second hypothesis is that the multiscale entropy (MSE) complexity index will show consistent test-retest reliability across both blocked and random testing groups when following clinical concussion management timelines.

Participants will complete five SOT sessions on the SMART Balance Master: three tests in one day with 20-minute breaks in between, followed by a test on day 45 and another on day 50.

DETAILED DESCRIPTION:
Understanding Sport-Related Concussion and Postural Stability Assessment

Over the past two decades, sport-related concussion (SRC) has gained significant attention from the media, as well as the medical and scientific communities. Despite this, SRC remains one of the most complex and least understood neurological injuries faced by sports medicine clinicians. Many physical activities, especially contact sports, pose a high risk of SRC due to direct or indirect impacts to the head, neck, face, or body, which can transmit force to the brain.

Research has consistently shown that contact sports have a high incidence of concussion, and various tools for assessing SRC have been developed. Baseline testing is a key component of concussion management, ideally conducted before the start of the sports season and before contact drills begin. It serves as a reference point for an athlete's pre-injury performance, making it easier to identify and manage SRC when an injury occurs. Recommended baseline testing includes neurocognitive assessments, balance tests, and symptom evaluations.

Postural stability assessments are widely used to evaluate concussed athletes by measuring coordination between motor and sensory functions. Balance deficits can indicate impaired integration of the visual, vestibular, and somatosensory systems, which are crucial for maintaining an upright posture. Researchers have explored both computerized dynamic posturography and clinical balance tests as part of SRC management protocols. These methods have been validated to detect subtle declines in balance performance, with both clinical and computerized balance assessments commonly used to monitor postural stability in athletes three to five days after a concussion.

The use of postural stability testing in SRC management is becoming more common among sports medicine clinicians. Clinical and laboratory-based balance evaluations are now routinely integrated into concussion protocols. One of the most advanced tools for assessing postural stability is the Sensory Organization Test (SOT), which is designed to identify balance impairments related to sensory and motor function coordination. The SOT, performed using the SMART Balance Master®, provides a more detailed assessment of balance function under various conditions. While computerized balance testing systems like the SMART Balance Master® are expensive and time-intensive, they offer more precise and objective data for concussion evaluation and recovery monitoring.

A. Challenges in Measuring Postural Stability

One common method for assessing postural stability is analyzing center of pressure (COP) data from the SMART Balance Master®. However, current approaches often rely on linear analysis, which may not fully capture the complexity of human movement. A widely used metric, the equilibrium score (ES), has three key limitations:

1. Variability in Individual Stability Limits - The ES calculation is based on a fixed range of motion (12.5° total: 8.0° anterior sway and 4.5° posterior sway). Since each individual's stability limits vary due to factors like age and height, using a standardized estimate can introduce errors.
2. Limited Data Utilization - The ES is derived from only two extreme sway angles, disregarding the full range of sway data. This simplification may overlook critical postural control details and allow different combinations of sway angles to produce identical ES values.
3. Exclusion of Biomechanical Factors - Important variables like body mass, height, and ankle torque, which influence postural stability, are not included in ES calculations. This omission raises concerns about the accuracy of the ES as a measure of balance control.

B. Advancing Postural Stability Analysis with Multiscale Entropy

To address these limitations, researchers have begun using entropy-based measures to analyze postural control. One such method, multiscale entropy (MSE), assesses the complexity of biological data across multiple time scales. Unlike traditional linear measures, MSE provides deeper insights into the regularity and adaptability of postural control during movement tasks.

MSE has shown promise in analyzing COP displacement more effectively than ES calculations. Since ES is derived from estimated sway angles rather than direct COP measurements, it may not capture the full complexity of postural control. By contrast, MSE considers fluctuations in COP over different time scales, offering a more comprehensive understanding of postural stability in athletes.

C. Establishing Reliability and Validity in SRC Assessment

Regardless of whether clinicians use ES or MSE for SRC assessment, two key issues must be addressed:

1. Practice Effects in Equilibrium Scores - Research on ES practice effects with repeated testing is limited. Establishing whether multiple test administrations influence ES values is crucial for obtaining valid baseline measurements. Eliminating practice effects ensures that changes in postural stability reflect genuine recovery rather than repeated exposure to testing.
2. Test-Retest Reliability of MSE and ES - No studies have examined the test- retest reliability of MSE and ES over clinically relevant concussion management timeframes. If MSE proves to be a more reliable metric, it could enhance SRC evaluation and improve return-to-play decision- making. Reliable assessment tools are essential for sports medicine clinicians when determining an athlete's readiness to safely return to competition after a concussion.

As SRC research continues to evolve, improving balance assessment methods is critical for enhancing concussion management. While ES remains a widely used measure, its limitations highlight the need for more sophisticated approaches like MSE. Establishing the reliability of both ES and MSE in SRC assessment will help refine concussion protocols and provide sports medicine clinicians with better tools for evaluating postural stability and recovery.

D. Normative Data and Influencing Factors in Postural Stability Assessment Normative data provide essential reference points for interpreting postural stability assessments in sport-related concussion (SRC) management. Studies examining balance performance across different populations have highlighted significant variations due to factors such as age, gender, and baseline stability levels. For instance, younger individuals typically demonstrate greater postural control compared to older adults, as age-related declines in sensory integration and musculoskeletal function affect balance. Additionally, gender differences in postural stability have been observed, with research suggesting that males and females may rely on different sensory inputs for maintaining equilibrium. Women, for example, may exhibit greater reliance on visual feedback, while men often depend more on proprioceptive and vestibular cues.

When interpreting equilibrium scores (ES) and multiscale entropy (MSE) values, it is crucial to consider how these normative variations influence test outcomes. Clinical assessment tools, such as the Sensory Organization Test (SOT)and center of pressure (COP) analyses, must account for these demographic differences to improve diagnostic accuracy and individualized concussion management. Moreover, balance performance can be influenced by an athlete's prior history of SRC, lower extremity injuries, and sport-specific training, further emphasizing the need for individualized baseline assessments.

Given these complexities, future research should establish age- and gender-specific normative datasets for postural stability assessments in athletes. By refining these reference values, clinicians can enhance their ability to detect post-concussion impairments and track recovery progress, ultimately leading to more precise return-to-play decisions.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-24
* Healthy young adults without balance problems

Exclusion Criteria:

* Self-reported history of concussion or head injury within the past 6 months
* Current musculoskeletal injuries in the lower extremities and/or other body parts that may affect postural stability
* Physical illnesses including visual or vestibular pathologies
* Consumption of any pharmacological substances affecting balance, recreational drugs, or alcoholic beverages within 24 hours prior to the balance test
* Self-reported severe tiredness or fatigue

Ages: 20 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteer college students without concussion
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2008-12-03 (Actual); Primary Completion 2011-12-31 (Actual); Study Completion 2014-04-16 (Actual)

PRIMARY OUTCOMES:
Practice effects: Serial Administration of the sensory organization test in health adults | From the time of enrollment until 60 days post-enrollment
  The Sensory Organization Test (SOT), administered using the SMART Balance Master®, generates one overall Composite Equilibrium Score (ES) and four sub-composite scores: somatosensory (SOM), visual (VIS), vestibular (VEST), and preference (PREF).
  The primary outcome measure will be the Composite ES, which reflects the overall balance performance and is expressed as a score ranging from 0 to 100, with higher scores indicating better balance. The sub-composite scores represent specific components of the balance system-somatosensory, visual, vestibular, and sensory integration preference-and are also scored on a scale from 0 to 100. Higher sub-composite scores similarly indicate better function in each respective domain.
  All scores are calculated by the software embedded within the SMART Balance Master® system. The Composite ES and sub-composite scores will be reported as the primary outcome measure to ensure consistency in units of measurement.
Test-Retest Reliability of the SOT using Mutlscal Entropy values and Equilibrium Scores in Heathy Adults | From the time of enrollment until 60 days post-enrollment
  The SMART Balance Master® provides a composite equilibrium score and four sub-composite scores (somatosensory, visual, vestibular, and preference), each ranging from 0 to 100, with higher scores indicating better balance performance.
  Additionally, Complexity Index (CI) scores are computed from raw center of pressure (COP) data exported from the SMART system and analyzed using MATLAB. CI, ranging from 0 to 20, quantifies postural complexity based on filtered COP data in the anterior-posterior and medial-lateral directions. Higher values indicate greater balance complexity.
  Although the outcomes involve two different units, this is not a concern, as the study focuses on test-retest reliability. Reliability coefficients (e.g., ICC) and standard error of measurement are unitless or interpreted within the context of each score type.

SECONDARY OUTCOMES:
Normative Sensory Organization Test and Multiscale Entropy Scores for Concussion Evaluation in a Healthy Young Population | From the time of enrollment until 60 days post-enrollment
  The Sensory Organization Test (SOT) on the SMART Balance Master® objectively quantifies postural stability deficits, producing a composite equilibrium score and four sensory-specific sub-scores, each ranging from 0 to 100. Higher scores reflect better balance performance.
  Additionally, the Complexity Index (CI) is calculated from raw center of pressure (COP) data exported from the SMART system and analyzed in MATLAB. CI values, ranging from 0 to 20, quantify postural complexity based on filtered COP signals in the anterior-posterior and medial-lateral directions, with higher values indicating greater complexity.
  Although SOT and CI use different measurement scales, this poses no issue, as the study's goal is to establish normative data for both metrics in healthy young adults. Given the limited normative data available for the SOT and the absence of published CI norms in this population, including both measures strengthens their utility for sports concussion assessment.

IPD SHARING:
Plan to Share IPD: No